CLINICAL TRIAL: NCT01720589
Title: Development of Rich & Creamy Melt® Organic Cooking Blend for Oxidative Stability and Reducing Childhood Obesity
Brief Title: Effect of Dietary Fat Cooking Blend on Energy Expenditure in Children
Acronym: Melt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Prosperity Organic Foods (Unknown); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Research Associate, St. Luke's-Roosevelt Hospital Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-33610-19482
Record Dates: First submitted 2012-10-17; First posted 2012-11-02 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Childhood Obesity
Keywords: Obesity; Dietary fat; Energy expenditure; Food intake
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Freezing; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melt (test oil) (Experimental): Participants will consume a muffin containing 20 g of dietary fat provided by the test oil and their energy expenditure will be measure post-prandially for 6 hours. At the end of the measurement period, participants will consume a cookie containing 10 g of fat provided by the test oil and their food intake at an ad libitum meal will be measured 1 hour later.
  Interventions: Dietary Supplement: Melt (test oil)
- Corn oil (control) (Active Comparator): Participants will consume a muffin containing 20 g of dietary fat provided by the control oil and their energy expenditure will be measure post-prandially for 6 hours. At the end of the measurement period, participants will consume a cookie containing 10 g of fat provided by the control oil and their food intake at an ad libitum meal will be measured 1 hour later.
  Interventions: Dietary Supplement: Corn oil (control)

INTERVENTIONS:
Dietary Supplement: Melt (test oil)
  Arms: Melt (test oil)
Dietary Supplement: Corn oil (control)
  Arms: Corn oil (control)

SUMMARY:
The purpose of this study is to test the effects of a cooking oil blend of dietary fats rich in medium chain triglycerides on energy expenditure and food intake in overweight and obese children.

ELIGIBILITY:
Inclusion Criteria:

* age 15-18
* body mass index 85% percentile or higher for age/sex
* weight stable

Exclusion Criteria:

* ±5 lbs weight change in the the 3 months prior
* use of medications
* dietary allergies
* metabolic disorder
* eating disorder
* behavioral or psychological disorders

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Thermic effect of food | 6 h
  Measurement of thermic effect of food over 6 hours after a meal rich in test oil and control oil. The thermic effect of food is the difference between post-prandial energy expenditure and basal energy expenditure. We will assess the difference in thermic effect of food over a 6-hour period between the test oil and the control oil.
Respiratory quotient/fat oxidation | 6 h
  Measurement of substrate oxidation by indirect calorimetry over 6 hours after consumption of the test oil and control oil. We will specifically calculate carbohydrate and fat oxidation rates over the 6-hour period post-prandially and compare rates of oxidation of these two substrates between the test oil and the control oil.
Food intake | single meal
  Measurement of food intake at a single meal served 1 hour after a pre-load containing 8-10 g of the test oil and the control oil

SECONDARY OUTCOMES:
Glucose | 6 h
  Measurement of glucose over 6 hours after consumption of the test oil and control oil
Feelings of appetite and satiety | 6 h
  Measurement of feelings of appetite and satiety by visual analog scales over 6 hours after consumption of the test oil and control oil
Insulin | 6 hours
  Measurement of insulin over 6 hours after consumption of the test oil and control oil
Leptin | 6 hours
  Measurement of leptin over 6 hours after consumption of the test oil and control oil
Ghrelin | 6 hours
  Measurement of ghrelin over 6 hours after consumption of the test oil and control oil
Peptide YY | 6 hours
  Measurement of peptide YY over 6 hours after consumption of the test oil and control oil
Glucagon like peptide 1 | 6 hours
  Measurement of glucagon like peptide 1 over 6 hours after consumption of the test oil and control oil

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — St. Luke's-Roosevelt Hospital Center; Cygnia Rapp, Principal Investigator — Prosperity Organic Foods
Locations (1):
- St. Luke's/Roosevelt Hospital, New York, New York, United States